CLINICAL TRIAL: NCT01681784
Title: Studies of Biomarkers in Different Urodynamic Diagnoses of Female Patients With Lower Urinary Tract Symptoms
Brief Title: Studies of Biomarkers in Female Lower Urinary Tract Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Professor Ho-Hsiung Lin, National Taiwan University Hospital
Other Study IDs: 200901031R
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2009-03

CONDITIONS: Disorder of the Lower Urinary Tract
Keywords: lower urinary tract symptoms; biomarkers; urodynamic studies
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients' voided urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine the sensitivity and specificity of urinary NGF, PGE2, IL-6, EGF or combinations in diagnosing different urodynamic diagnoses.

DETAILED DESCRIPTION:
Abstract

Background/Purpose:

Urodyamic study is an objective method to evaluate female patients with lower urinary tract symptoms (LUTS). However, this method includes place a urinary catheter, thus prevents it as a routine method to evaluate and follow up patients with LUTS. Therefore, it is necessary to find a simple and objective method to help in evaluating female patients with LUTS. Several kinds of biomarker had been reported in diagnosing patients with overactive bladder; however, the sensitivity remained poor. The aim of this study is to find a useful biomarker, biomarkers, or combinations, with the aid of urodynamic study, to objectively and precisely in evaluating the female patients with LUTS.

Patients and Methods:

We will perform a prospective study to recruit 300 female patients with LUTS at the outpatient clinic of Department of Obstetrics and Gynecology of National Taiwan University Hospital and Far Eastern Memorial Hospital.

All patients will be asked to complete OABSS, UDI-6 & IIQ-7 questionnaires, voiding diary, 20-min pad test and urodynamic studies. Urinary nerve growth factor, prostaglandin E2, interleukin-6 and epidermal growth factor were also measured. Besides, we will also recruit 30 female patients without LUTS in our outpatient clinic, and they will be asked to complete the above questionnaire and examinations except pad test and urodynamic studies.

Possible Results:

With the comparison of the above parameters between non-LUTS and LUTS patients, we can answer the questions that (1) the mean values of urinary NGF, PGE2, IL-6, EGF in different urodynamic studies, (2) the sensitivity and specificity of urinary NGF, PGE2, IL-6, EGF or combinations in diagnosing different urodynamic diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with lower urinary tract symptoms

Exclusion Criteria:

* acute cystitis

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with lower urinary tract symptoms and underwent urodynamic studies
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan